CLINICAL TRIAL: NCT06086964
Title: Effect of Therapeutic Diet Along With Special Physiotherapy Program on Growth Motor Development and Cognitive Function in Autism Spectrum Children
Brief Title: Effect of Therapeutic Diet With Physiotherapy on Gross Motor and Cognition of Autistic Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Jazan (Other Government)
Responsible Party: Principal Investigator, Mohamed Moustafa Mohamed Ahmed, assistant professor of basic science, physical therapy department, University of Jazan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: HAPO-10-Z-001
Record Dates: First submitted 2023-10-10; First posted 2023-10-17 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Autistic Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder | interventions — Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group A (Experimental): 15 autistic child will receive gluten and casein free diet.
  Interventions: Other: therapeutic diet.
- Group B (Experimental): 15 autistic child will receive physical therapy program.
  Interventions: Other: physiotherapy
- Group C (Experimental): 15 autistic child will receive combination of gluten and casein free diet with physical therapy program.
  Interventions: Other: therapeutic diet.; Other: physiotherapy
- Group D (No Intervention): the group of no intervention as a control group.

INTERVENTIONS:
Other: therapeutic diet. — gluten and casein free diet.
  Arms: Group A; Group C
Other: physiotherapy — specific physiotherapy developmental program according to the pre evaluation of gross motor status.
  Arms: Group B; Group C

SUMMARY:
: A clinical trial will be conducted to investigate the effect of free-gluten/ casein diet along with specific physiotherapy program on gross motor development and cognitive function in 3-12 years old children with ASD, And thus establish a streamlining of nutrition and physical activity for children with autism and ASD.

DETAILED DESCRIPTION:
Autism is a complex neurological and developmental disability that appears within early developmental stages of life. Autism affects the normal functioning of the brain, communication development as well as social skills of the child. Autism has been regarded as a life-long condition and it cannot be cured. However, severity may decrease through special diet and physiotherapy program.

In Saudi Arabia, the prevalence revealed that confirmed cases of ASD were 42,500, and many remained undiagnosed A target group of (60) children diagnosed with autism or ASD, attending the paediatric psychiatry outpatient clinic and autism centres will be enrolled in this clinical trial study, which will be conducted in Jazan City-Saudi Arabia.

The inclusion criteria will be as follows: (1) parental consent, (2) age 3-12 years, and (3) a diagnosis of autism or ASD. Exclusion criteria were as follows: (1) autism associated with a genetic syndrome, (2) patients with comorbidities (3) known food allergy leading to avoidance of certain foods, and (4) mother or primary caretaker not available to be adherent to the prescribed diet. Three groups will be designed: (1) autistic children with regular diet and physiotherapy program. (2) Autistic children on free gluten/casein diet and (3) Autistic children on free gluten/casein diet and subjected to specific physiotherapy program. The study will be continued for 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Children diagnosed with autism spectrum disorders.
* GMFCs 4

Exclusion Criteria:

* autistic children with any musculoskeletal deformities.
* autistic children with any bulbar affection lead to problem in swallowing.

Ages: 3 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 2023-10-17 (Actual); Primary Completion 2024-02-16 (Actual); Study Completion 2024-03-12 (Actual)

PRIMARY OUTCOMES:
gross motor development | 2 hours
  Bruininks-oseretsky test of motor proficiency-1
Cognitive function | 2 hours
  using Bimet IQ test

CONTACTS AND LOCATIONS:
Locations (1):
- Jazan University, Jizan, Gizan, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No
after finishing we can share the data with request.